CLINICAL TRIAL: NCT00315081
Title: Therapy With Bromocriptine in Patients With Symptomatic Risperidone-Induced Hyperprolactinemia
Brief Title: Risperidone-Induced Hyperprolactinemia Treated With Bromocriptine
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University Hospital, Bonn (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 150-05
Record Dates: First submitted 2006-04-13; First posted 2006-04-17 (Estimated); Last update posted 2006-04-17 (Estimated); Status verified 2005-11

CONDITIONS: Schizophrenia; Hyperprolactinemia
Keywords: Schizophrenia; Hyperprolactinemia; Risperidone; Bromocriptin
MeSH Terms: conditions — Schizophrenia; Hyperprolactinemia | interventions — Bromocriptine

INTERVENTIONS:
Drug: Bromocriptin

SUMMARY:
Antipsychotic drugs can cause a clinically relevant hyperprolactinemia due to blocking the dopamine receptors in the pituitary.Schizophrenic patients suffering from a neuroleptic-induced hyperprolactinemia will be examined endocrinologically. Adverse drug effects and diagnoses will be confirmed by measuring hormones.

DETAILED DESCRIPTION:
Antipsychotic drugs can cause a clinically relevant hyperprolactinemia due to blocking the dopamine receptors in the pituitary.Depending on its concentration hyperprolactinemia causes a median hypogonadism with estrogen insufficiency in women and testosterone insufficiency in men by inhibiting the pulsatile GnRH-secretion.The hyperprolactinemia-induced symptoms have been successfully medicated for years with dopamine agonists like bromocriptine.

In patients with psychiatric diseases hyperprolactinemia is usually not treated with dopamine agonist fearing a reexacerbation of the underline psychiatric disease. In a few studies and casuistically the treatment of neuroleptic-induced hyperprolactinemia with bromocriptine has been shown to be effective without causing reexacerbation of psychotic symptoms.

Schizophrenic patients suffering from a neuroleptic-induced hyperprolactinemia (in extremis galactorrhoea and amenorrhoea. in women, loss of libido and erectile dysfunction in men) will be examined endocrinologically. Adverse drug effects and diagnoses will be confirmed by measuring hormones (prolactin, LH, FSH, testosterone, estradiol). In case of a clear symptomatic, neuroleptic-induced hyperprolactinemia patients will be medicated with bromocriptin. Therapeutical success will be determined endocrinologically in week 0, 1, 2, 3, 4, 8, 12, 16, 20 and 24 together with a psychiatric examination (PANSS, HAM-D, Simpson-Angus Scale (SAS)). Safety of therapy will be ensured by the close meshed psychiatric examinations.

ELIGIBILITY:
Inclusion Criteria:

* Female and male schizophrenic patients.
* Antipsychotic treatment with risperidone.
* Diagnosis of a clinically relevant hyperprolactinemia.
* No indication of disturbance of the somato-, cortico or thyreotropic hypophysis-axis (IGF-1, cortisol, ACTH, TSH, FT3, FT4)

Exclusion Criteria:

* Severe somatic disease, especially coronary disease.
* Acute psychotic exacerbation.
* Pregnancy

Ages: 18 Years to 60 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20
Dates: Start 2006-05; Study Completion 2008-05

PRIMARY OUTCOMES:
Prolactin
LH
FSH
Testosterone
Estradiol

SECONDARY OUTCOMES:
PANSS
HAM-D
Simpson Angus Scale (SAS)

CONTACTS AND LOCATIONS:
Overall Officials: Wolfgang Maier, MD, Principal Investigator — University of Bonn, Department of Psychiatry
Locations (1):
- University of Bonn, Department of Psychiatry, Bonn, Northrhine-Westfalia, Germany

REFERENCES:
- [Background] Bliesener N, Yokusoglu H, Quednow BB, Klingmuller D, Kuhn KU. Usefulness of bromocriptine in the treatment of amisulpride-induced hyperprolactinemia: a case report. Pharmacopsychiatry. 2004 Jul;37(4):189-91. doi: 10.1055/s-2004-827176. No abstract available. PMID 15467977